CLINICAL TRIAL: NCT00984490
Title: Pre-Surgical Trial of Metformin in Patients With Operable Breast Cancer
Brief Title: Metformin Hydrochloride in Treating Women With Stage I or Stage II Breast Cancer That Can Be Removed By Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow accrual
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Vandana Abramson, Professor of Medicine, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC BRE 0942; P30CA068485 (NIH); VU-VICC-BRE-0942
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Results first posted 2012-07-13 (Estimated); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metformin (Experimental): Metformin: 850 mg orally (PO) twice daily (BID) for 7-21 days, discontinued 24-36 hrs prior to surgery
  Interventions: Drug: metformin hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: metformin hydrochloride — Metformin: 850 mg orally (PO) twice daily (BID) for 7-21 days, discontinued 24-36 hrs prior to surgery
Other: laboratory biomarker analysis — Blood and tissue collection to determine the in situ biologic effect of metformin

SUMMARY:
RATIONALE: Metformin hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I trial is studying how well metformin hydrochloride works in treating women with stage I or stage II breast cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the in situ effects of metformin hydrochloride on proliferation (Ki67) and apoptosis (caspase-3) in women with operable stage I or II breast cancer.

Secondary

* To determine the in situ biologic effect of metformin hydrochloride on the AMP kinase, MTOR/PI3K, and IGF pathways in breast cancer (tissue S6K and phospho S6K, p53, p63, and p73 levels as well as p53 [(Ser-15), if wild-type p53 is present], p63 [Ser-66/68, Ser-301, and Ser-361], and p73 [Y-99] phosphorylation, PTEN [clone 6H2.1], phospho-Akt [S473], insulin receptor substrate 1 and 2 [IRS-1 and IRS-2], and LKB1).
* To determine if molecular classification (basal-type vs luminal A vs luminal B) and the established p63 and p73 RNA microarray gene signatures correlate with the metformin hydrochloride-induced effects on proliferation (Ki67), apoptosis (caspase-3) and the selected biomarkers (listed above) in breast cancer.
* To collect and analyze pre- and post-treatment peripheral blood specimens for serum glucose and insulin levels, as well as circulating IGF-1 and IGF binding protein 3 (IGFBP3).

OUTLINE: Patients receive oral metformin hydrochloride twice daily for 7-21 days. Approximately 24-36 hours after the last dose of metformin hydrochloride, patients undergo surgical resection (total mastectomy or segmental resection with lymph node evaluation) of tumor.

Patients undergo blood and tissue sample collection periodically for biomarker analysis.

ELIGIBILITY:
Inclusion:

* Patients must provide informed written consent
* Eastern Cooperative Oncology Group performance status 0-1.
* Clinical stage I, II or IIIA invasive mammary carcinoma, any estrogen receptors(ER), progesterone receptors (PR), or Human Epidermal Growth Factor Receptor (HER2/NEU) status
* Patients who have measurable residual tumor at the primary site Measurable disease: a mass that can be reproducibly measured by physical examination and/or ultrasound and is at least 1 cm in size by physical examination or ultra-sound measurement
* Patients who will undergo surgical treatment with either segmental resection or total mastectomy with lymph node evaluation
* Consultations: All patients should be evaluated by a surgeon prior to study entry.
* Available core biopsies from the time of diagnosis. These may include sections paraffin-embedded material.
* Female subjects ≥18 years of age
* No prior chemotherapy for this primary breast cancer.
* Patients with a prior history of contralateral breast cancer are eligible if they have no evidence of recurrence of their initial primary breast cancer.
* Women may have been taking tamoxifen or raloxifene as a preventive agent prior to study entry but must have discontinued the drug for at least 21 days prior to study enrollment.
* Patients must have adequate hepatic and renal function. All tests must be obtained less than 4 weeks from study entry. This includes:
* Creatinine </= to 1.5X upper limits of normal
* Bilirubin, SGOT, SGPT < or = to 1.5X upper limits of normal
* Able to swallow and retain oral medication

Exclusion:

* Patients with locally advanced disease who are candidates and wish to undergo preoperative chemotherapy at the time of initial evaluation. Patients with operable locally advanced disease (stage IIIA) are eligible for participation.
* Locally recurrent breast cancer
* Evidence of distant metastatic disease (i.e. lung, liver, bone, brain, etc.)
* History of diabetes mellitus
* Pregnant or lactating women
* Metformin treatment within 30 days of study entry
* Serious medical illness that in the judgment of the treating physician places the patient at high risk of operative mortality.
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel. Subjects with ulcerative colitis are also excluded.
* History of other malignancy. Subjects who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinomas are eligible
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
* History of a medical condition leading to chronic hypoxemia and/or ischemia (congestive heart failure, emphysema or chronic lung disease requiring supplemental oxygen)
* Chronic metabolic acidosis (serum HCO3- < or = to 20 or requiring sodium bicarbonate supplementation)
* Concurrent anti-cancer therapy (chemotherapy, radiotherapy, immunotherapy, hormonal therapy, or any other biologic therapy)
* Concurrent treatment with an investigational agent
* Use of an investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the first dose of study drug.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-09; Primary Completion 2010-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Mayer, M.D., Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Emory University Hospital, Atlanta, Georgia
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited patients from September 24, 2009 through June 28, 2011.
Pre-assignment Details: Five patients enrolled on this study during the first nine months. Accrual continued to be slow causing its premature closing.
Groups:
- Metformin: Metformin: 850 mg PO twice a day for 7-21 days (discontinued 24-36 hrs prior to surgery
Period: Overall Study
Arm/Group | Metformin
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Metformin
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Ki67 Levels Before and After Treatment
Description: Change in Ki67 levels in pre-treatment, pre-surgery and post-treatment, surgically excised breast tissue. Measured by percentage of positive-staining nuclei with a minimum of 0% to a maximum of 100%. A mean score is determined.
Time Frame: baseline and between 8-23 days
Population: No Ki67 levels were determined. This clinical trial was closed due to slow accrual
Groups:
- Metformin: Metformin: 850 mg orally (PO) twice a day for 7-21 days, discontinued 24-36 hrs prior to surgery
Arm/Group | Metformin
Number analyzed (Participants) | 0

2. Secondary Outcome: Changes in Circulating Insulin-like Growth Factor 1 (IGF-1) and IGF Binding Protein 3 (IGFBP-3)
Description: Effect of study drug on circulating IGF-1 and IGFBP-3 as measured in ng/mL in peripheral blood samples taken pre-treatment and post-treatment with metformin
Time Frame: baseline and 23 days
Population: No levels of IGF-1 and IGFBP-3 were determined. This clinical trial was closed due to slow accrual.
Groups:
- Metformin: Metformin: 850 mg PO twice a day for 7-21 days (discontinued 24-36 hrs prior to surgery)
Arm/Group | Metformin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Metformin
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 4/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=5)
diarrhea (Gastrointestinal disorders) | 4 (5)
nausea (Gastrointestinal disorders) | 2 (2)
vomiting (Injury, poisoning and procedural complications) | 1 (1)
weight loss (Investigations) | 1 (1)

LIMITATIONS AND CAVEATS:
Because this study was closed prematurely, no assay level markers or pathways were performed consequently no data are available to provide results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes